CLINICAL TRIAL: NCT04183075
Title: Clinical Trial to Assess the Impact of a Nutritional Supplement on the Recovery of the Nutritional Status of Elderly Patients With Spontaneous Hip Fracture
Brief Title: Impact of a Nutritional Supplement on the Recovery of the Nutritional Status of Patients With Spontaneous Hip Fracture
Acronym: IRENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratorios Ordesa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRENE
Record Dates: First submitted 2019-11-25; First posted 2019-12-03 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Hip Fractures; Malnutrition
Keywords: phase angle; nutritional supplement
MeSH Terms: conditions — Hip Fractures; Malnutrition | interventions — Carbohydrates; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FontActiv Superprotein/Hypercaloric Fiber (Experimental): Full Nutritional Supplement
  Interventions: Dietary Supplement: FontActiv Superprotein/Hypercaloric Fiber
- Carbohydrates and C Vitamin (Active Comparator): Nutritional Supplement
  Interventions: Dietary Supplement: Carbohydrates and C Vitamin

INTERVENTIONS:
Dietary Supplement: FontActiv Superprotein/Hypercaloric Fiber — The product under study has a liquid presentation, in 200 ml bottles, ready to take
  Arms: FontActiv Superprotein/Hypercaloric Fiber
Dietary Supplement: Carbohydrates and C Vitamin — The control product will be prepared with equal presentation and taste as similar as possible tan study product
  Arms: Carbohydrates and C Vitamin

SUMMARY:
Multicenter, prospective, randomized, double-blind, interventional study with a nutritional supplement against placebo in a cohort of patients hospitalized for hip fracture.

DETAILED DESCRIPTION:
Hip fracture is a very prevalent pathology in the elderly population. It is estimated that 35-40% of people over 65 suffer a drop per year, and above 75 years this percentage is even higher, with hip fractures being one of the most serious consequences.With regard to malnutrition, the investigators know that aging carries an increased risk of suffering from decreased appetite and intake and changes in body composition. According to different series, the percentage of malnutrition in patients with hip fracture ranges from 13% to 60%. According to the hospital protocols in Spain in elderly people with spontaneous hip fracture, it is important to perform a nutritional screening during the first 24-48 hours of admission, to evaluate their nutritional status and apply a dietary treatment.

The IRENE study aims to determine whether phase angle and reactance, measured by electrical bioimpedance by vector analysis (BIVA) are related to functional recovery in patients with hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years old.
* Patients admitted to hospital by spontaneous hip fracture and requiring surgery.
* Patients who after hip intervention are included in rehabilitation protocols with outpatient rehabilitation plan.
* Patients who agree to participate by signing informed consent or their regular caregivers grant consent.

Exclusion Criteria:

* Patients who have a hip fracture from high-impact trauma or secondary to bone pathology (such as neoplasm).
* Patients with concomitant diseases such as severe hepatic impairment, severe renal impairment, insulin-dependent diabetes melitus and decompensated diabetes mellitus.
* Patients who require clinical stabilization before surgery beyond 72 hours.
* Patients receiving emergency surgery.
* Patients with previous prostheses.
* Patients with pacemakers.
* Patients who are not likely to complete the follow-up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Compare changes in nutritional status between groups based on phase angle | From baseline to month 4
  Compare changes in nutritional status between patients taking nutritional supplement under study and control group based on phase angle measurement (morphological criterion)
Compare changes in nutritional status between groups based on force measurement | From baseline to month 4
  Compare changes in nutritional status between patients taking nutritional supplement under study and control group based on force measurement using hand-grip strength ( functional criteria).

SECONDARY OUTCOMES:
To compare functional recovery | From baseline to month 4
  Compare functional recovery using the Barthel Scale between patients taking nutritional supplement under study and placebo. It is scored on a scale ranging from 0 to 100, with 90 being the maximum score if the patient is in a wheelchair.
To compare the morphological recovery by muscle ultrasound | From baseline to month 4
  Compare the morphological recovery valued by muscle ultrasound between patients taking nutritional supplement under study and placebo. Ultrasound performed at baseline and month 4
To compare changes in Mini Nutrition Assessment test for aged people | From baseline to month 4
  Compare changes in the Mini Nutrition Assessment score between the two study groups. This is a validated test for aged people to assess the nutritional status. Good nutritional state: more than 17points. Bad nutritional state: less than 17 points.
To compare the evolution of the Global Subjective Valuation questionnaire | From baseline to month 4
  To compare the evolution of the Global Subjective Valuation between the two study groups. It is a method designed to estimate nutritional status through medical history and physical examination. Each of the sections is valued as mild, moderate or severe, being severe the worst nutritional condition.
Compare changes between groups in the Charlson index | From baseline to month 4
  Charlson index takes into account the number and severity of accompanying diseases to predict the risk of death. Each pathology that patient has, has a number. The higher the number, the worst prediction.
Number of participants that have to be readmitted at the hospital. | From baseline to month 4
  Compare the difference in hospital re-admissions between the two study groups.
Number of participants that die during the study | From baseline to month 4
  Compare the differences in mortality within four months of the start of the study between the two study groups
Compare changes in the ratio RCP/Prealbumin index in the blood analysis | From baseline to month 4
  Compare changes in the ratio RCP/Prealbumin index between the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Manuel Garcia Almeida, Principal Investigator — Hospital Clínico de Málaga
Locations (2):
- Spain (2):
  - Hospital Clínico de Málaga, Málaga, Andalusia
  - Hospital Virgen del Rocío, Seville, Andalusia